CLINICAL TRIAL: NCT02488395
Title: Superior Colliculus Activity in Parkinson Disease: a Potential Marker? fMRI Brain Activation in Response to Visual Stimuli.
Brief Title: Superior Colliculus Activity in Parkinson Disease: a Potential Marker?
Acronym: AGIRPARK
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C14-58; IDRCB (Registry Identifier: 2014-A01835-42)
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2021-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Non-motor symptoms; Visual deficits; Superior colliculus; fMRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- de novo Parkinson's patients: This group includes de novo Parkinson's patients who have just been diagnosed and not started their treatment at the inclusion.
  This group will perform three fMRI sessions at different crucial steps of their normal follow up with a neurologist. Their visual abilities will be tested with an ophthalmologic evaluation and their sensitivity to contrast with a visual psycho-physics test.
  Interventions: Other: fMRI; Other: Ophthalmologic evaluation; Other: visual psychophysics test
- matching controls: This group includes age-matching control participants to the first Parkinson group.
  This group will perform one fMRI session. Their visual abilities will be tested with an ophthalmologic evaluation and their sensitivity to contrast with a visual psycho-physics test.
  Interventions: Other: fMRI; Other: Ophthalmologic evaluation; Other: visual psychophysics test

INTERVENTIONS:
Other: fMRI — The investigators will use a non invasive fMRI technique centred on the superior colliculus during the presentation of flickered check-boards with varying contrast (1, 3, 5 and 9 %).
Other: Ophthalmologic evaluation — The aim of this experiment is the evaluate the functional state of a visual structure. Therefore, with this ophthalmologic test, the investigators will control if the participant does not present major visual deficits. This examination will evaluate the visual acuity and the visual field. A funduscopic examination will also be performed to check the retina.
Other: visual psychophysics test — This test will allow to control the sensitivity of the participant to our contrast. The participant will be asked to look at screen on which three static check-boards will be presented. The participant will have to choose the two check-boards with the closest contrast.

SUMMARY:
The ultimate goal of this project is to evaluate a possible new strategy to diagnose earlier Parkinson's disease, using the superior colliculus as a biomarker.

Preliminary data from the investigator's group in a rat model of Parkinson's disease suggest that the superior colliculus, a sensory structure, show an early deficit in visual processing. The investigator's data also suggests that with the evolution of the disease, this structure presents a neuronal re-organisation leading which causes a sensory rebound after the introduction of the treatment. The light responses in the superior colliculus were faster, bigger in amplitude and lasted longer (Rolland et al., 2012). Those results raise an important question about the superior colliculus functional state in Parkinson's patients. If this structure have a similar neuroplasticity, the investigators could hypothesize that the superior colliculus may also present a sensory rebound when introducing the treatment. If this hypothesis is true, the accelerated and amplified light responses of this structure may explain the difficulties felt by the patients to inhibit reflexive saccades induced by the appearance of unexpected visual stimuli. Indeed, the superior colliculus is involved in the orientation of the head and eye toward any sudden changes in our environment (Wurtz and Albano, 1980) and the light responses of this structure are strongly correlated with the speed of the saccade (Marino et al., 2012).

Therefore, the investigators want to test if a similar deficit could be observed in the superior colliculus of newly diagnosed PD patients. Data will be compared to matching controls.

DETAILED DESCRIPTION:
This project aims at better understanding the physiopathology of Parkinson's disease and the effect of the administration of the classical medical treatment. The main aim of this project is to evaluate the possibility of an early detection using a new original strategy. The investigators want to demonstrate the predictive value of the superior colliculus light responses as an early biomarker.

The investigators will perform functional magnetic resonance imagery (fMRI) to measure the BOLD light responses of the superior colliculus at different key stages of the normal medical follow up of Parkinson's patients by the neurologist (when diagnosed, when introducing the first treatment and when the treatment is stabilised).

Two groups of participants will be tested: a) a group of de novo patients, which have just been diagnosed and haven't started their treatment; b) a group of matching controls.

A first fMRI session (S1) will be performed to compare the light induced BOLD response of the superior colliculus between de novo patients and their matching controls. This session will evaluate a possible visual processing dysfunction in the superior colliculus of newly diagnosed patients.

Parkinson's patients will then start their treatment and a second session (S2) will be done on this group shortly after the introduction of the treatment to measure its acute effect. If the superior colliculus of those patients presents a sensory rebound, the investigators should observe a bigger light-induced BOLD response after the treatment compared to before the treatment.

A third session (S3) will be performed after the optimal adjustment of the treatment on motor symptoms which would be around six month after the start of the treatment. This adjustment is long and difficult, realized by the neurologist according to its effect on the motor symptoms. Those two last fMRI will allow the investigators to compare the effect of the introduction of the treatment on the motor symptoms, known to not improve correctly at this stage, and on non-motor symptoms (visual processing deficits in this project) from which no information are available to the investigators knowledge.

ELIGIBILITY:
Inclusion Criteria:

* De novo parkinson's patients being just diagnosed (stage 1 according to the Hoehn and Yahr scale: first unilateral signs with no discomfort in everyday life) without a current dopaminergic treatment and who have not started their anti-parkinsonian treatment.
* Both Parkinson's patients and their age matching control must not present a major visual pathology (mainly in the retina) which may interfere with the visual task.
* Signed informed and free consent.
* Matching controls must not present a neurological or psychiatric troubles.
* For the matching controls: There are no contraindication on current treatments apart from those to treat other neurological disease than Parkinson's disease or psychiatric troubles.
* For Parkinson's patients: There are no contraindication on current treatments apart from those to treat neurological troubles including anti-parkinsonian treatment, or psychiatric troubles.
* As a precaution, the investigators will check that no MRI exam has been performed during the week preceding our fMRI.

Exclusion Criteria:

* Parkinson's patients with important tremor limiting the validity of the fMRI acquisition.
* Adult under supervision
* Incapacity to understand the consent explanations.
* Impossibility to participate to the whole experimental protocol.
* No affiliation to a health insurance.
* Consent not signed by a participant or refusal by the participant to participate to the experiment.
* Pregnancy or breast feeding woman.
* Administrative or justice freedom restricted participant.

Exclusion Criteria specific for MRI:

* Pacemaker, neurosensorial stimulator or implanted defibrillator.
* Presence of ocular or cerebral ferromagnetic material.
* Respiratory disease (i.e. asthma), cardio-vascular deficits, claustrophobia

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Groups of de novo Parkinson's patients and their age matching controls.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Light responses measure in the superior colliculus | 2 hours / session

CONTACTS AND LOCATIONS:
Overall Officials: Elena Moro, MD/PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Michel Dojat, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (3):
- France (3):
  - CHU de Grenoble, Grenoble, Isere
  - Grenoble Institute of Neurosciences, Grenoble, Isere
  - IRMAGE, Grenoble, Isere

REFERENCES:
- [Result] Bellot E, Kauffmann L, Coizet V, Meoni S, Moro E, Dojat M. Effective connectivity in subcortical visual structures in de novo Patients with Parkinson's Disease. Neuroimage Clin. 2022;33:102906. doi: 10.1016/j.nicl.2021.102906. Epub 2021 Dec 7. PMID 34891045
- [Result] Moro E, Bellot E, Meoni S, Pelissier P, Hera R, Dojat M, Coizet V; Superior Colliculus Study Group. Visual Dysfunction of the Superior Colliculus in De Novo Parkinsonian Patients. Ann Neurol. 2020 Apr;87(4):533-546. doi: 10.1002/ana.25696. Epub 2020 Feb 19. PMID 32030799